CLINICAL TRIAL: NCT01950078
Title: The Possible Correlations Between the Genes Related to Pain Sensation and the Pain Sensitivity in the General Population
Status: Completed | Type: Observational
Sponsor: Xianwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: Gene and Pain
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pain; Surgery
Keywords: gene polymorphism; pain perception; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Heparin anti-coagulated blood (5 ml) was collected from the periphery venous of subjects and all blood samples were stored at -80℃. Genomic DNA was extracted from the blood samples using a guanidinium isothiocyanate method.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- surgical patients: grouped by receiving surgery
- Healthy volunteers group: grouped by healthy college students

SUMMARY:
Objective: This study was conducted to explore the possible correlation between some gene related to pain sensation and individual basal pain perception and postoperative pain intensity in the general population. Methods: Patients receiving elective surgery under general anesthesia were recruited into this study. The investigators measured their preoperative pressure pain threshold (PPT) and pressure pain tolerance (PTO). Pain intensity at rest and movement after the operation was evaluated . And the PCA drug consumption were recorded. Also there were healthy college students volunteer be recruited into this study. The investigators measured their experimental pain sensitivity including pressure pain threshold (PPT) and pressure pain tolerance (PTO), etc. Then genotyping was carried out.

DETAILED DESCRIPTION:
Subjects with the following diseases were excluded: known history of chronic disease, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or drug abuse, heavy smoker, Pregnancy or at lactation period .

ELIGIBILITY:
Inclusion Criteria:

* •Aged 18-65 years

  * Receiving elective gynecological laparoscopic surgery
  * Anesthesiologists (ASA) physical status I or II
  * Agreed to participate the research

Exclusion Criteria:

* •History of chronic pain

  * Psychiatric diseases
  * Diabetes mellitus
  * Severe cardiovascular diseases
  * Kidney or liver diseases
  * Alcohol or drug abuse
  * Heavy smoker
  * Pregnancy or at lactation period
  * Disagree to participate to the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anticipative 500 healthy volunteers and 1000 surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 1533 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, MD, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Patients | Healthy Volunteers Group
Started | 1025 | 508
Completed | 1005 | 496
Not Completed | 20 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Patients | Healthy Volunteers Group | Total
Number analyzed (Participants) | 1005 | 496 | 1501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 7 | 18
  Between 18 and 65 years | 990 | 489 | 1479
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1005 | 309 | 1314
  Male | 0 | 187 | 187
Region of Enrollment [Number; unit: participants]
  China | 1005 | 496 | 1501

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Pressure Pain Threshold (PPT)
Description: The probe of pressure algometer was positioned perpendicularly to the skin surface of the patient, and the investigator applied continuous pressure at approximately the same rate according to the visual LCD display on the algometer. subjects were asked to say "pain" when they started to feel pain during the stimulation. The value from the LCD was recorded as the pressure pain threshold.
Time Frame: 30 minutes before the operation
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Surgical Patients | Healthy Volunteers Group
Number analyzed (Participants) | 1005 | 496
kg/cm2 | 2.33 (0.97) | 3.24 (1.25)

2. Secondary Outcome: Preoperative Pressure Pain Tolerance (PTO)
Description: The probe of pressure algometer was positioned perpendicularly to the skin surface of the patient, and the investigator applied continuous pressure at approximately the same rate according to the visual LCD display on the algometer. subjects were asked to say "ok" when they started to feel the pain became intolerable during the stimulation. The value from the LCD was recorded as the pressure pain tolerance.
Time Frame: 30 minutes before the operation
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Surgical Patients | Healthy Volunteers Group
Number analyzed (Participants) | 1005 | 496
kg/cm2 | 4.65 (1.66) | 6.38 (2.56)

ADVERSE EVENTS:
Arm/Group | Surgical Patients | Healthy Volunteers Group
Serious Adverse Events (participants affected / at risk) | 0/1005 | 0/496
Other Adverse Events (participants affected / at risk) | 0/1005 | 0/496

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes